CLINICAL TRIAL: NCT02154035
Title: Quantitative Measurement and Correlates of the Latent HIV Reservoir in Virally Suppressed Ugandans
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914123; 14-I-N123
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-26

CONDITIONS: HIV
Keywords: Viral Suppression; Functional Cure; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: HIV-infected patients on ART with suppressed viral loads, defined as <40 copies per ml over a period of 10-18 months.
- Group 2: HIV-infected patients on ART with suppressed viral loads, defined as <40 copies per ml over a period of 10-18 months.

SUMMARY:
Background:

Human Immunodeficiency Virus (HIV) is the virus that causes AIDS. HIV can hide in the blood for many years, even in people who have their HIV infection under control. HIV that is hiding in the blood is called the "latent HIV reservoir." Researchers want to find out more about it in this study. This knowledge may help them develop new ways to prevent or control HIV. This study will draw its participants from the Rakai Health Sciences Program in rural southwestern Uganda.

Objective:

- To measure and learn about the latent HIV reservoir in Ugandans with HIV.

Eligibility:

- Men and women at least 18 years of age with HIV.

Design:

* Participants will have a medical history and physical exam. Their medical records will be reviewed. Researchers will ask participants about their health and recent illnesses. Participants able to get pregnant will have their urine tested for pregnancy.
* Participants will have their finger pricked to see if they have enough red blood cells to be eligible for the study.
* If eligible, participants will have blood drawn through a needle in the arm. Their blood will also be tested for other diseases.
* After the blood draw, participants will be asked to stay seated or lying down if they are not feeling well for up to 30 minutes.

DETAILED DESCRIPTION:
Despite prolonged antiretroviral therapy (ART), HIV-1 can persist as transcriptionally inactive proviruses in resting memory CD4+T cells. This latent reservoir has a long half-life, and is believed to be the largest impediment to a cure by ART alone. The latent reservoir may be established when activated CD4+ T cells become infected and subsequently revert back to a resting memory state. A major approach to eradicating HIV-1 involves reversing latency in patients on ART. Cells harboring induced proviruses could be lysed by HIV-1-specific cytolytic T lymphocytes, while ART blocks new rounds of infection. The descriptions of the "Berlin patient" and "Mississippi baby" suggest that a functional cure for HIV is possible. This has led to an expansion of research examining HIV latency in the context of sustained viral suppression with an eye towards developing a possible cure regimen that could be used on a large scale. However, it has recently been demonstrated that the latent HIV reservoir could be 60 times larger than previously believed. The recent report that two HIV patients receiving CCR5competent bone marrow transplants had a reemergence of circulating HIV after fully suppressive therapy was discontinued suggests that a functional cure for large groups of individuals will continue to be an elusive goal.

The vast majority of HIV-infected individuals currently live in sub-Saharan Africa where fully suppressive ART is expanding rapidly. Due to this expansion, a large number of Africans will be eligible candidates for cure treatment when one comes available. However, strategies needed to establish a functional cure may differ in African populations due to differences in endemic infectious disease load and in cellular immune activation among Africans as compared to Western populations. To date, there have been no systematic studies to quantify the latent reservoir in HIV-infected Africans. This is a longitudinal, descriptive study to measure the size of the latent HIV reservoir in virally suppressed HIV infected individuals residing in Uganda and to examine the immunological and virologic correlates of the latent reservoir. The study will draw its participants from a National Institutes of Health (NIH) International Center for Excellence in Research (ICER) site, located at the Rakai Health Sciences Program (RHSP) in rural southwestern Uganda. One group of subjects will be comprised of 70 HIV-infected patients who are on ART with suppressed viral loads <40 copies per ml over a period of 10-18 months. A second group includes 20 individuals with a known window of seroconversion (an HIV-negative test result no more than 18 months before the first HIV-positive test result). A third group will be comprised of 10 HIV infected subjects with suppressed viral load <40 copies per ml over a period of 10-18 months, while not on ART. A fourth group will include 30 individuals living with HIV on ART with suppressed viral loads, who have known windows of seroconversion, and initiated ART early. Study participation will require a visit with a fingerstick hemoglobin screening and a blood draw, once a year for a period of 20 years. Plasma and cells from the blood will be separated and processed for quantitative viral latency, viral clonality analysis, circulating cytokine and chemokine analysis, co-culture, and flow cytometric and serologic assays for selected immunological parameters. Viral latency results and clonality measurements will be compared within each individual for changes in the reservoir size and make-up that might occur over 20 years of continual viral suppression in order to calculate the T1/2 or decay rate of the total latent reservoir and it s component proviral populations. Samples collected from individuals with known infection dates will be used to estimate the formation curve of the latent reservoir. Overall reservoir size and decay and formation rates will be interpreted in relation to values previously collected from HIV-infected individuals in the United States.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 18 years of age
  2. Hemoglobin >11g/dL as assessed by fingerstick rapid test
  3. Weight >40 kilograms
  4. A historical diagnosis of HIV infection as indicated by any positive serological test (ELISA, HIV rapid test, or Western Blot)
  5. Virally suppressed as defined as at least two historical viral loads <40 copies/ml obtained between 10-18 months apart, and no intervening detectable viral load result >= 40 copies/ml obtained during this period
  6. Most recent historical viral load result obtained within a year prior to the screening visit
  7. Willingness to undergo genetic testing

EXCLUSION CRITERIA:

1. Women who are pregnant will be excluded as the required blood draw may cause anemia and because of perturbations due to hormonal or immunosuppressive states that could impact the reservoir.
2. Inability to follow study instructions or to provide informed consent
3. Any condition deemed by the investigators to be a contraindication to study participation including active, serious infections (other than HIV infection) during the 2 weeks prior to enrollment.
4. Malignancies of any kind (e.g., Kaposi's sarcoma)
5. Therapy with systemic steroids, immunosuppressants or immunomodulating agents
6. Coagulation defects or other serious bleeding disorders
7. Current use of medications which could affect clotting.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will draw its participants from an NIH International Center for Excellence in Research (ICER) site, located at the Rakai Health Sciences Program (RHSP) in rural southwestern Uganda. Since 1994, over 12,000 adults aged 15-49 years of age have been under annual surveillance in an open cohort, the Rakai Community Cohort Study (RCCS). Within the RCCS, the Rakai Program has conducted multiple observational, basic science, behavioral and operations research studies, and has conducted complex community and individual randomized HIV and sexually transmitted disease (STD) prevention trials.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-05-31; Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Explore the level of immune activation in virally suppressed HIV-infected Africans in correlation with the size of the reservoir | Enrollment
  Explore the level of immune activation in virally suppressed HIV-infected Africans in correlation with the size of the reservoir
Examine and measure the levels of latent HIV reservoirs in virally suppressed Ugandans and compare to that observed in Western (US) cohorts | Enrollment
  Examine and measure the levels of latent HIV reservoirs in virally suppressed Ugandans and compare to that observed in Western (US) cohorts
Determine the role of endemic infectious diseases, nadir CD4 count, and length of fully suppressive therapy on latent HIV reservoir size | Enrollment
  Determine the role of endemic infectious diseases, nadir CD4 count, and length of fully suppressive therapy on latent HIV reservoir size
Evaluate in vitro potential latency reversal agents. | Enrollment
  Evaluate in vitro potential latency reversal agents.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Rakai Health Sciences Program Uganda Virus Research Institute, Kalisizo, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho YC, Shan L, Hosmane NN, Wang J, Laskey SB, Rosenbloom DI, Lai J, Blankson JN, Siliciano JD, Siliciano RF. Replication-competent noninduced proviruses in the latent reservoir increase barrier to HIV-1 cure. Cell. 2013 Oct 24;155(3):540-51. doi: 10.1016/j.cell.2013.09.020. Epub 2013 Oct 24. PMID 24243014
- [Background] Wightman F, Ellenberg P, Churchill M, Lewin SR. HDAC inhibitors in HIV. Immunol Cell Biol. 2012 Jan;90(1):47-54. doi: 10.1038/icb.2011.95. Epub 2011 Nov 15. PMID 22083528